CLINICAL TRIAL: NCT00614861
Title: A Clinical Survey on Satisfaction of Pain Management in Patients With Non-cancer Pain in Taiwan
Brief Title: Pain Satisfaction Survey
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CR014659
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Pain
Keywords: Non-cancer pain; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 001
  Interventions: Other: Non-cancer pain management survey

INTERVENTIONS:
Other: Non-cancer pain management survey — Non-cancer pain management survey

SUMMARY:
The purpose of this study is to survey pain management satisfaction in patients with non-cancer pain.

DETAILED DESCRIPTION:
This is a multi-center, Observational study consisting of a one time survey to assess pain management satisfaction for patients with non-cancer pain. The purpose of this study is to develop a large clinical database for the results of the pain management satisfaction questionnaire. All information collected from hospitals will be used to evaluate patient satisfaction of pain management and to improve the quality of life for patients with non-cancer pain Observational study - No study drug administered

ELIGIBILITY:
Inclusion Criteria:

* Patients who have visited out patient department (OPD) and who are actively treated for pain

Exclusion Criteria:

* Patients with cancer pain
* Patients with known or suspected psychotic disease or mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have visited out patient department (OPD) who are treated actively for pain
Sampling Method: Probability Sample
Enrollment: 2929 (Actual)
Dates: Start 2007-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To explore pain management satisfaction in patients with non-cancer pain in Taiwan. | Visit 1

SECONDARY OUTCOMES:
To collect the information about Quality of Life in patients with non-cancer pain | Visit1
To collect information about medication for pain management | Visit1

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd